CLINICAL TRIAL: NCT05590208
Title: Sleeve Gastrectomy With Cruroplasty and Omental Rape for Treatment of Morbid Obesity With Reflux Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, assistant professor of general surgery, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fac.med 22.64
Record Dates: First submitted 2022-10-01; First posted 2022-10-21 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2022-12

CONDITIONS: Obesity, Morbid; GERD
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sleeve gastrectomy+ cruroplasty + omental rape (Experimental): sleeve gastrectomy+ cruroplasty + omental rape
  Interventions: Procedure: sleeve gastrectomy+ cruroplasty+ omental rap

INTERVENTIONS:
Procedure: sleeve gastrectomy+ cruroplasty+ omental rap — sleeve gastrectomy+ cruroplasty+ omental rap

SUMMARY:
in this study the investigators will test anew technique to mange patients with morbid obesity and GERD by doing sleeve gastrectomy plus cruroplasty and omental rape around the gastroesophageal junction

DETAILED DESCRIPTION:
in this study the patients that have morbid obesity concomitant GERD will managed by sleeve gastrectomy plus cruroplasty then stripe from the momentum is fashioned and is raped around the gastroesophageal junction

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 60
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
the effect on GERD | 6 months
  change in GERD symptoms using either upper GIT endoscopy or GERDQ questionnaire

SECONDARY OUTCOMES:
weight loss | 12 months
  the effect on weight loss determined by percentage of excess weight loss, percentage of total weight loss and change of BMI
comorbidities | 12 months
  change in comorbidities including diabetes by change in hemoglobin C level, hypertension by measuring arterial blood pressure using sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Minia university hospital, Minya, Egypt